CLINICAL TRIAL: NCT03442829
Title: Impact of Repeated Sweet Breakfasts on Subsequent Sweet Food Preferences and Intakes
Brief Title: Repeated Sweet Breakfasts and Subsequent Sweet Food Preferences and Intakes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Collaborators: University of Bristol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: KAPR2018
Record Dates: First submitted 2018-02-01; First posted 2018-02-22 (Actual); Results first posted 2020-08-27 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Repeated Sweet Food Consumption
Keywords: sweet taste, food preferences, food intake
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Intervention allocation will be undertaken by a researcher not directly involved with participants following randomization by drawing lots.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sweet food consumption (Experimental): Sweet breakfasts. Participants are asked to consume a sweet breakfast every day for three weeks (excepting on three days when outcomes will be assessed (days 0, 7 and 21, day 21 reported). All foods will be provided.
  Interventions: Behavioral: Sweet food consumption
- Non-sweet food consumption (Active Comparator): Non-sweet breakfasts. Participants are asked to consume a non-sweet breakfast every day for three weeks (excepting on three days when outcomes will be assessed (days 0, 7 and 21, day 21 reported). All foods will be provided.
  Interventions: Behavioral: Non-sweet food consumption

INTERVENTIONS:
Behavioral: Sweet food consumption — Sweet food consumption at breakfast
  Arms: Sweet food consumption
Behavioral: Non-sweet food consumption — Non-sweet food consumption at breakfast
  Arms: Non-sweet food consumption

SUMMARY:
This study will assess the impact of repeated sweet breakfast consumption versus repeated non-sweet breakfast consumption on subsequent sweet and non-sweet food preferences and intakes

DETAILED DESCRIPTION:
Participants will be randomized to receive either sweet or non-sweet breakfasts for three consecutive weeks, and impacts on food preferences and intakes will be assessed at baseline (day 0), after 1 week (day 7), and after three weeks (day 21). Preferences for sweet and non-sweet foods will be assessed during two taste tests at each assessment time, where six different foods will be rated. Sweet and non-sweet food consumption will also be measured at two meals at each assessment time - breakfast and lunch. Identical buffet meals composed of sweet and non-sweet foods suitable for consumption at breakfast and lunch will be provided ad-libitum. Intervention breakfasts will only be consumed on the days between test days.

ELIGIBILITY:
Inclusion Criteria:

* No known food allergy
* No known taste or appetite abnormalities
* Non-smoker
* Habitually eats breakfast
* Able to provide consent and complete all study measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Appleton, PhD, Principal Investigator — Bournemouth University, UK; Peter Rogers, PhD, Principal Investigator — University of Bristol
Locations (1):
- Bournemouth University, Bournemouth, US and Canada Only, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The full study protocol is currently available from the PI on reasonable request. All generated data will be available from the PI, following completion and publication of the work on reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available following completion and publication of the study. Data will be stored for ten years following publication of the work.
Access Criteria: Direct contact and reasonable request of the PI.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sweet Food Consumption: Sweet breakfasts. Participants are asked to consume a sweet breakfast every day. All foods will be provided.
  Sweet food consumption: Sweet food consumption at breakfast
- Non-sweet Food Consumption: Non-sweet breakfasts. Participants are asked to consume a non-sweet breakfast every day. All foods will be provided.
  Non-sweet food consumption: Non-sweet food consumption at breakfast
Period: Overall Study
Arm/Group | Sweet Food Consumption | Non-sweet Food Consumption
Started | 27 | 27
Completed | 23 | 25
Not Completed | 4 | 2
Not completed — Scheduling clash | 3 | 1
Not completed — Illness unrelated to study | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sweet Food Consumption | Non-sweet Food Consumption | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.2 (7.0) | 23.5 (4.4) | 23.9 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 9 | 9 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 27 | 27 | 54
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.0 (3.9) | 23.2 (3.2) | 23.6 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Food Preferences
Description: Ratings of three sweet and three non-sweet foods during a taste test at breakfast. Ratings measured using 100mm VAS scales for different hedonic factors - pleasure, sweetness, desire to eat). Scores range from 0-100 where 0=least and 100=greatest for each hedonic factor. Assessments made on Day 0, 7 and 21, Day 21 reported.
Time Frame: 3 weeks from baseline
Population: Intention-to-Treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Sweet Food Consumption | Non-sweet Food Consumption
Number analyzed (Participants) | 27 | 27
units on a scale
  Sweet foods | 73 (3.1) | 68 (4.0)
  Non-sweet foods | 54 (3.6) | 50 (3.8)

2. Primary Outcome: Food Intake
Description: Amount of sweet and non-sweet foods consumed during breakfast on test days (days 0, 7 and 21, day 21 reported)
Time Frame: 3 weeks from baseline
Population: Intention-to-Treat
Measure: Mean (Standard Error); unit: percentage of total food consumed
Arm/Group | Sweet Food Consumption | Non-sweet Food Consumption
Number analyzed (Participants) | 27 | 27
percentage of total food consumed
  Percent weight consumed from sweet foods | 28.5 (3) | 36 (4)
  Percent energy consumed from sweet foods | 37 (4) | 39 (4)

3. Secondary Outcome: Hunger Ratings
Description: Ratings of subjective perceptions (two meals). Ratings measured using 100mm VAS scales for different subjective factors - hunger, thirst, fullness. Scores range from 0-100 where 0=least and 100=greatest for each subjective factor. Assessments made on Day 0, 7 and 21, Day 21 reported.
Time Frame: 3 weeks from baseline
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sweet Food Consumption | Non-sweet Food Consumption
Number analyzed (Participants) | 27 | 27
units on a scale
  Hunger | 72 (19) | 68 (24)
  Fullness | 15 (11) | 20 (30)
  Thirst | 65 (30) | 67 (27)

4. Secondary Outcome: Food Preferences at Lunch
Description: Ratings of three sweet and three non-sweet foods during a taste test at lunch. Measures are the same as those used at breakfast. Ratings measured using 100mm VAS scales for different hedonic factors - pleasure, sweetness, desire to eat). Scores range from 0-100 where 0=least and 100=greatest for each hedonic factor. Assessments made on Day 0, 7 and 21, Day 21 reported.
Time Frame: 3 weeks from baseline
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sweet Food Consumption | Non-sweet Food Consumption
Number analyzed (Participants) | 27 | 27
units on a scale
  Sweet foods | 70 (15) | 67 (21)
  Non-sweet foods | 54 (21) | 52 (18)

5. Secondary Outcome: Food Intake at Lunch
Description: Amount of sweet and non-sweet foods consumed during lunch on test days (days 0, 7 and 21, day 21 reported).
Time Frame: 3 weeks from baseline
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: percentage of total food consumed
Arm/Group | Sweet Food Consumption | Non-sweet Food Consumption
Number analyzed (Participants) | 27 | 27
percentage of total food consumed
  Percent weight consumed from sweet foods | 27 (17) | 32 (19)
  Percent energy consumed from sweet foods | 33 (17) | 37 (22)

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: verbal self-report
Arm/Group | Sweet Food Consumption | Non-sweet Food Consumption
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT03442829/Prot_SAP_000.pdf